CLINICAL TRIAL: NCT06528028
Title: Relationship Between Different Administration Regimens of Ceftazidime/Avibactam and Clinical Outcomes in Patients With Severe Infection: a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Relationship Between Different Administration Regimens of Ceftazidime/Avibactam and Clinical Outcomes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH3420202401
Record Dates: First submitted 2024-07-10; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-06

CONDITIONS: Anti-Infective Agent
Keywords: Anti-Infective Agent

STUDY DESIGN:
Intervention Model Description: Treatment group and control group
Masking Description: A non-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Ceftazidime/avibactam（Taidingping®, Qilu Pharmaceutical Co., Ltd.） loading dose of 2.5g (2h infusion), then the standard dose and administration schedule, namely 2.5gQ8h, continuous infusion, the dose can be adjusted according to the instructions of renal function，The duration of medication is determined by the clinician
  Interventions: Drug: CAZ/AVI
- control group (Experimental): Ceftazidime/avibactam（Taidingping®, Qilu Pharmaceutical Co., Ltd.）were given a load dose of 2.5g (2h infusion), followed by 2.5gQ8h, the dose can be adjusted according to renal function.The duration of medication is determined by the clinician.
  Interventions: Drug: CAZ/AVI

INTERVENTIONS:
Drug: CAZ/AVI — continuous infusion is used
  Other Names: Continous group
  Arms: treatment group
Drug: CAZ/AVI — 2h-infusion is used
  Other Names: Intermittent group
  Arms: control group

SUMMARY:
Ceftazidime/avibactam (CAZ/AVI) is a new β-lactam drug, which has good antibacterial effect against carbapenem resistant enterobacter. However, previous studies found that CAZ/AVI had a low PK/PD compliance rate after the recommended dose of the drug instructions.Therefore, this study was intended to explore the clinical efficacy of different administration schedules of CAZ/AVI for patients with severe infection, and further analyze the correlation between CAZ/AVI PK/PD parameters and clinical efficacy and adverse reactions.

DETAILED DESCRIPTION:
1. Main purpose The main objective of this study was to verify that the clinical efficacy of treatment group (load dose of 2.5g, then continuous infusion of 2.5gQ8h, the dose can be adjusted according to renal function) with severe infection was superior to that of the control group (standard dose and administration regimen of ceftazidime/avibactam, i.e. 2.5gQ8h, 2h infusion).Dose can be adjusted according to renal function).
2. Secondary purpose (1) To investigate the relationship between different administration regimens and bacterial clearance and 28-d mortality (2) To explore the correlation between different dosing regimens and PK/PD compliance rate (3) To explore the correlation between different administration regimens and adverse drug reactions

ELIGIBILITY:
Inclusion Criteria:

Multiple-resistant negative bacteria Sensitive to ceftazidime/avibactam Received intravenous infusion of ceftazidime/avibactam

Exclusion Criteria:

Allergic to ceftazidime/avibactam Blood sample not be collected Pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Clinical effective rate | 14 days
  According to the Technical Guidelines for Clinical Trials of Antimicrobial Drugs, clinical efficacy is defined as: (1) effective: symptoms, signs, pathogenic microbiology and various tests and examination indicators are significantly improved;(2) Ineffective: the patient's condition has not improved or worsened, and other antibacterial drugs need to be replaced.Effective rate = Number of effective cases/total cases x 100%.

SECONDARY OUTCOMES:
Bacterial removal | 14 days
  Defined as clearance or change of existing bacteria within two weeks of medication.
28-d mortality | 28 days
  Defined as whether a patient died at 28-d after follow-up.28-d Mortality rate = Number of deaths/group size x 100%.
PK/PD compliance rate | 14 days
  PK/PD compliance rate = number of qualified persons/number of groups × 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Xu, Ph.D, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Intensive Care Unit, Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No